CLINICAL TRIAL: NCT04204720
Title: A Comparison of Intravascular Injection With Chiba Needle and Whitacre Needle During Caudal Epidural Block : a Prospective Study
Brief Title: A Comparison of Intravascular Injection With Chiba Needle and Whitacre Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-06-007
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Spinal Stenosis Lumbar; Disk Herniated Lumbar
MeSH Terms: interventions — Needles

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Whitacre (Active Comparator): Group whitacre receives the whitacre needle during caudal block
  Interventions: Device: needle (Whitacre)
- Group Chiba (Experimental): Group chiba receives the chiba needle during caudal block
  Interventions: Device: needle (Chiba)

INTERVENTIONS:
Device: needle (Chiba) — intravascular injection using chiba needle during caudal epidural block
  Arms: Group Chiba
Device: needle (Whitacre) — intravascular injection using whitacre needle during caudal epidural block
  Arms: Group Whitacre

SUMMARY:
Caudal epidural injection (CEI) is effective for spinal pain. However, intravascular injection may occur during CEI, which can lead to hematoma, neurologic deficit and local anesthetics systemic toxicity. Whitacre type needle has been reported to be effective for reducing intravascular injection during transforaminal epidural injection. In this study, we compared the Chiba needle and Whitacre needle on incidence of intravascular injection during CEI.

DETAILED DESCRIPTION:
A total of 164 caudal epidural injections were performed in patients with disc herniation or spinal stenosis on lumbosacral region. Patients were randomly allocated to Group Whitacre (n=82) and Group Chiba (n=82). Patients in Group Whitacre received caudal epidural injection using Whitacre type needle and those in Group Chiba received the procedure using Chiba type needle. Intravascular injection was assessed with blood aspiration and angiography during real-time fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients with low back pain and/or leg radicular pain under diagnoses as disc herniation or spinal stenosis

Exclusion Criteria:

* allergy to local anesthetics or contrast medium, coagulopathy, local infection at the injection site, and systemic infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
incidence of intravascular injection | 5 minute
  incidence of intravascular injection during caudal block

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No